CLINICAL TRIAL: NCT06133608
Title: The Effect of Mobilization Training on Kinesiophobia and Fear of Falling in Patients Undergoing Hip Arthroplasty After Femur Fracture
Brief Title: Kinesiophobia and Fear of Falling After Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, MAHİNUR DURMUŞ İSKENDER, Assistant Professor, Kastamonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuU2
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Fear of Other Medical Care
Keywords: Fear of moving; Fear of falling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients in the intervention group will be educated by watching videos on the first day after surgery, in addition to routine clinical education. On the 10th post-operative day, the patients will be called by the researcher and the "Tampa Kinesiophobia Scale" and "Fall Activity Scale" will be administered.
  Interventions: Other: MOBILIZATION TRAINING
- Control (No Intervention): The control group will receive routine clinical training. On the 10th post-operative day, the patients will be called by the researcher, and the "Tampa Kinesiophobia Scale" and "Fall Activity Scale" will be administered.

INTERVENTIONS:
Other: MOBILIZATION TRAINING — Things to consider in the hospital in the early period after surgery: The first day in the hospital after surgery, the importance of the abduction pillow and early mobilization,
  * Exercises performed in bed in the early period after surgery: Exercises such as ankle pump, ankle rotation, bed-supported knee bending, hip contraction, opening exercise, thigh exercise, straight leg raise,
  * Early standing up: Activities such as sitting in bed or on a chair, standing up with the help of a walker, walking,
  * Exercises performed while standing: Exercises such as lifting the knee, opening the leg to the side,
  * Daily living activities: It will provide information on regulating ADLs such as bathing, dressing, using the toilet, getting into and driving the car, going up and down stairs, eating, sleeping, doing housework, sexual life, and information about the safety precautions that should be taken at home.
  Arms: Experimental

SUMMARY:
This study will be conducted as intervention research to determine the effect of mobilization training to be provided to the patient undergoing hip arthroplasty on postoperative kinesiophobia and fear of falling. The project will be carried out with 50 voluntary patients (25 intervention, 25 control) aged over 65 who came to Hospital for hip arthroplasty after femur fracture, can communicate, have no advanced sensory loss related to vision and hearing, do not have a psychiatric history, and will undergo hip arthroplasty surgery for the first time. Data will be collected using a "Sociodemographic Characteristics Questionnaire", the "Tampa Scale for Kinesiophobia", and "the Fall Activity Scale". Appropriate statistical methods will be used in the analysis of the data. Patients in the control group will be given routine care during the study. Patients in the experimental group will receive technology-assisted mobilization training in addition to routine care. Before mobilization, a training video loaded into a tablet will be given to patients. Written permission will be taken from the ethics committee and the institution for the implementation of the research and written consent will be obtained from the patients.

DETAILED DESCRIPTION:
As a result of the changes that occur in old age, individuals face different problems and risks more frequently than the younger age group. One of the most important among these is falls, which cause high mortality and morbidity in this age group. Hip fractures that occur after a fall are the most distressing injuries that elderly individuals experience. Hip arthroplasty is one of the treatment methods preferred by patients who have hip fractures after a fall. After hip arthroplasty, elderly patients may avoid mobilization due to the fear of falling and damaging the prosthesis. This can lead to restriction of activities and a decrease in functional independence. This avoidance behavior increases with the fear of falling. Avoidance of movement due to fear of falling is defined as "kinesiophobia". Studies have stated that mobilization training before or after hip arthroplasty surgery is effective in postoperative mobilization. For this reason, it is thought that providing mobilization training to patients undergoing hip arthroplasty surgery will lead to more success in mobilization.

This study will be conducted as intervention research to determine the effect of mobilization training to be provided to the patient undergoing hip arthroplasty on postoperative kinesiophobia and fear of falling. The project will be carried out with 50 voluntary patients (25 intervention, 25 control) aged over 65 who came to Hospital for hip arthroplasty after femur fracture, can communicate, have no advanced sensory loss related to vision and hearing, do not have a psychiatric history, and will undergo hip arthroplasty surgery for the first time. Data will be collected using a "Sociodemographic Characteristics Questionnaire", the "Tampa Scale for Kinesiophobia", and "the Fall Activity Scale". Appropriate statistical methods will be used in the analysis of the data. Patients in the control group will be given routine care during the study. Patients in the experimental group will receive technology-assisted mobilization training in addition to routine care. Before mobilization, a training video loaded into a tablet will be given to patients. Written permission will be taken from the ethics committee and the institution for the implementation of the research and written consent will be obtained from the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo hip prosthesis due to femur fracture after a fall,
* Patients who were mobilized before falling,
* Being over 65 years of age
* Volunteering to participate in the research
* No previous hip arthroplasty
* Ability to read and write
* There is no perception disorder or psychiatric disorder that would hinder communication.

Exclusion Criteria:

* Having difficulty in communicating
* Severe sensory loss related to vision and hearing

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-06-05 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia | 10 days
  Tampa Scale for Kinesiophobia is a 17-question checklist and is used for acute and chronic low back pain, fibromyalgia, and diseases associated with musculoskeletal injuries and whiplash. A 4-point Likert scoring (1 = Strongly disagree, 4 = Completely agree) is used in the scale. A total score is calculated after reversing items 4, 8, 12 and 16. The person receives a total score between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia. Permission was obtained from the researchers for the use of the scale.

IPD SHARING:
Plan to Share IPD: No